CLINICAL TRIAL: NCT02853929
Title: Immunogenicity and Safety Study of a Booster Dose of GSK Biologicals' Infanrix Hexa™ (217744) in Healthy Infants Born to Mothers Vaccinated With Boostrix™ During Pregnancy or Immediately Post-delivery
Brief Title: Evaluation of Immunogenicity and Safety of a Booster Dose of Infanrix Hexa™ in Healthy Infants Born to Mothers Vaccinated With Boostrix™ During Pregnancy or Immediately Post-delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201334; 2014-001120-30 (EudraCT Number)
Record Dates: First submitted 2016-07-14; First posted 2016-08-03 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Diphtheria; Hepatitis B; Acellular Pertussis; Haemophilus Influenzae Type b; Tetanus; Poliomyelitis; Diphtheria-Tetanus-aPertussis-Hepatitis B-Poliomyelitis-Haemophilus Influenzae Type b Vaccines
Keywords: Pertussis; Immunogenicity; Poliomyelitis; Tetanus; Hepatitis B; Diptheria
MeSH Terms: conditions — Diphtheria; Hepatitis B; Haemophilus Infections; Tetanus; Poliomyelitis; Whooping Cough | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTpa Group (Experimental): This group will consist of healthy male or female infants, aged 9 months at the time of enrollment, born to mothers who received a single dose of Boostrix during pregnancy and a dose of placebo immediately post-delivery. All enrolled subjects in this group who will come back for subsequent visit will receive a booster dose of Infanrix hexa co-administered with Prevenar 13 according to the routine national/local immunization or study procedure
  Interventions: Biological: Infanrix hexa
- Control Group (Active Comparator): This group will consist of healthy male or female infants, aged 9 months at the time of enrollment, born to mothers who received a dose of placebo during pregnancy and single dose of Boostrix immediately post-delivery. All enrolled subjects in this group who will come back for subsequent visit will receive a booster dose of Infanrix hexa co-administered with Prevenar 13 according to the routine national/local immunization or study procedure
  Interventions: Biological: Infanrix hexa

INTERVENTIONS:
Biological: Infanrix hexa — All subjects will receive Infanrix hexa co-administered with Prevenar13 as a booster dose.

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of the Infanrix hexa booster dose given at 11-18 months of age to infants who received primary vaccination at 6-14 weeks. All infants in this booster study were born to pregnant women who participated in the study 116945 [DTPA (BOOSTRIX)-047] and having received the full primary vaccination series as per protocol requirement in study 201330 [DTPA (BOOSTRIX)-048.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally acceptable representatives (LAR(s)) who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* A male or female child 9 months of age at the time of enrolment.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects born to mothers who were vaccinated in 116945 [DTPA (BOOSTRIX)-047] study and having completed their primary vaccination series as per protocol requirement in study 201330 [DTPA (BOOSTRIX)-048 PRI].

Exclusion Criteria:

* Child in care
* Concurrently participating in another clinical study, within three months prior to the booster vaccine dose and at any time during the present booster study, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period within six months prior to the booster vaccine dose. For corticosteroids, this will mean prednisone ≥0.5mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* A vaccine not foreseen by the study protocol administered during the period starting from 30 days before the booster dose of study vaccine and ending 30 days after*, with the exception of inactivated influenza vaccine and other vaccines given as a part of the national/regional immunization schedule, that are allowed at any time during the study period.

  * In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its SPC or Product Information (PI) and according to the local governmental recommendations and provided a written approval of the Sponsor is obtained.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Major congenital defects.
* Serious chronic illness.
* Administration of immunoglobulins and/or any blood products during the period within three months before the booster dose of study vaccines or planned administration during the study period.
* Encephalopathy defined as an acute, severe central nervous system disorder occurring within 7 days following vaccination with Infanrix hexa and generally consisting of major alterations in consciousness, unresponsiveness, generalised or focal seizures that persist more than a few hours, with failure to recover within 24 hours.
* History of Hib, diphtheria, tetanus, pertussis, pneumococcal, poliovirus and hepatitis B diseases since the conclusion visit of study 201330 [DTPA (BOOSTRIX)-048 PRI].
* Previous booster vaccination against Hib, diphtheria, tetanus, pertussis, pneumococcus, hepatitis B and/or poliovirus since the conclusion visit of study 201330 [DTPA (BOOSTRIX)-048 PRI].
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines (e.g: antigen, excipients).
* Hypersensitivity to latex.
* History of any neurological disorders or seizures.
* Any condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Acute disease and/or fever at the time of vaccination.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.

Ages: 9 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 551 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- GSK Investigational Site, Carlton, Victoria, Australia
- Canada (3):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava - Vitkovice
  - GSK Investigational Site, Prague
- Finland (5):
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Novara, Piedmont
- Spain (9):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Móstoles
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Martinon-Torres F, Halperin SA, Nolan T, Tapiero B, Perrett KP, de la Cueva IS, Garcia-Sicilia J, Stranak Z, Vanderkooi OG, Kosina P, Rumlarova S, Virta M, Arribas JMM, Miranda-Valdivieso M, Novas BA, Bozensky J, Ortega MJC, Amador JTR, Baca M, Palomino EE, Zuccotti GV, Janota J, Marchisio PG, Kostanyan L, Meyer N, Ceregido MA, Cheuvart B, Kuriyakose SO, Mesaros N. Impact of maternal diphtheria-tetanus-acellular pertussis vaccination on pertussis booster immune responses in toddlers: Follow-up of a randomized trial. Vaccine. 2021 Mar 12;39(11):1598-1608. doi: 10.1016/j.vaccine.2021.02.001. Epub 2021 Feb 19. PMID 33612341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled in the study were infants aged 9 months at the time of enrollment, born to mothers vaccinated with Boostrix in study 116945 BOOSTRIX-047 [NCT02377349] and who received primary vaccination Infanrix hexa co-administered with Prevenar 13 in study 201330 BOOSTRIX-048 [NCT0242264]
Pre-assignment Details: 551 subjects were enrolled in this trial, out of which 540 received the booster dose of Infanrix hexa co-administered with Prevenar 13.
  11 subjects did not receive booster vaccination even though subject number had been allocated.
Groups:
- dTpa Group: This group included healthy male or female infants, aged 9 months at the time of enrollment, born to mothers who received a single dose of Boostrix during pregnancy and a dose of placebo immediately post-delivery.
  All enrolled subjects in this group who came back for subsequent visit received a booster dose of Infanrix hexa co-administered with Prevenar 13 according to the routine national/local immunization or study procedure
- Control Group: This group included healthy male or female infants, aged 9 months at the time of enrollment, born to mothers who received a dose of placebo during pregnancy and single dose of Boostrix immediately post-delivery.
  All enrolled subjects in this group who came back for subsequent visit received a booster dose of Infanrix hexa co-administered with Prevenar 13 according to the routine national/local immunization or study procedure
Period: Overall Study
Arm/Group | dTpa Group | Control Group
Started (Number of subjects enrolled) | 270 | 281
Vaccinated | 263 | 277
Completed | 259 | 277
Not Completed | 11 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subjects enrolled but not vaccinated | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dTpa Group | Control Group | Total
Number analyzed (Participants) | 270 | 281 | 551
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 270 | 281 | 551
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 128 | 255
  Male | 143 | 153 | 296
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 4 | 9 | 13
  Asian - East Asian Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 2 | 0 | 2
  White - Arabic / North African Heritage | 1 | 3 | 4
  White - Caucasian / European Heritage | 246 | 262 | 508
  Other | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Anti-diphtheria (Anti-D), Anti-tetanus (Anti-T), Anti-hepatitis B (Anti-HBs), Anti-poliovirus Type 1, Anti-poliovirus Type 2, Anti-poliovirus Type 3 and Anti-polyribosyl-ribitol Phosphate (Anti-PRP)
Description: Seroprotected subjects were defined as subjects with antibody concentrations/titres above or equal (≥) the assay cut-offs that are accepted immunological correlates of protection.
  0.1 International units per milliliter (IU/ml) for anti-D and anti-T, 10 milli-International units per milliliter (mIU/mL) for anti-HB's, 8 Effective Dose 50 (ED50) for anti-polio virus (type 1,2,3) and 0.15 microgram/milliliter (µg/mL) for anti-PRP were considered as immunological correlates of protection.
Time Frame: At one month after the booster dose (Day 30)
Population: Analysis was performed on the According to Protocol (ATP) cohort for immunogenicity, which included all subjects who met eligibility criteria, received the booster dose of the study vaccines and for whom assay results were available for antibodies against at least one study vaccine antigen component, after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 221 | 247
Participants
  Anti-D | 221 | 247
  Anti-T | 221 | 247
  Anti-HBs: number analyzed (Participants) | 216 | 241
  Anti-HBs | 215 | 239
  Anti-polio 1: number analyzed (Participants) | 204 | 228
  Anti-polio 1 | 204 | 228
  Anti-polio 2: number analyzed (Participants) | 201 | 227
  Anti-polio 2 | 201 | 227
  Anti-polio 3: number analyzed (Participants) | 188 | 210
  Anti-polio 3 | 188 | 210
  Anti-PRP | 221 | 246

2. Primary Outcome: Number of Subjects With a Booster Response to Pertussis Antigens (Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN))
Description: Booster response to PT, FHA and PRN antigens was defined as:
  * for subjects with pre-vaccination antibody concentration below the assay cut-off, post-vaccination antibody concentration ≥ 4 times the assay cut-off,
  * for subjects with pre-vaccination antibody concentration between the assay cut-off and below 4 times the assay cut-off, post-vaccination antibody concentration ≥ 4 times the pre-vaccination antibody concentration, and
  * for subjects with pre-vaccination antibody concentration ≥ 4 times the assay cut-off, post-vaccination antibody concentration ≥ 2 times the pre-vaccination antibody concentration
  Seronegative (S-) subjects are those who have antibody concentration less than (<) assay cut-off.
  Seropositive (S+) subjects are those who have antibody concentration ≥ assay cut-off prior to vaccination.
  Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti- FHA and 2.187 IU/mL for anti-PRN
Time Frame: At one month after the booster dose (Day 30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 215 | 241
Participants
  Anti-PT, S-: number analyzed (Participants) | 67 | 42
  Anti-PT, S- | 62 | 40
  Anti-PT, S+ (< 4*assay cut-off): number analyzed (Participants) | 108 | 126
  Anti-PT, S+ (< 4*assay cut-off) | 98 | 124
  Anti-PT, S+ (≥ 4*assay cut-off): number analyzed (Participants) | 40 | 73
  Anti-PT, S+ (≥ 4*assay cut-off) | 38 | 71
  Anti-PT, Overall | 198 | 235
  Anti-FHA, S-: number analyzed (Participants) | 8 | 3
  Anti-FHA, S- | 8 | 3
  Anti-FHA, S+ (< 4*assay cut-off): number analyzed (Participants) | 84 | 58
  Anti-FHA, S+ (< 4*assay cut-off) | 83 | 58
  Anti-FHA, S+ (≥ 4*assay cut-off): number analyzed (Participants) | 123 | 180
  Anti-FHA, S+ (≥ 4*assay cut-off) | 117 | 172
  Anti-FHA, Overall | 208 | 233
  Anti-PRN, S-: number analyzed (Participants) | 35 | 31
  Anti-PRN, S- | 34 | 31
  Anti-PRN, S+ (< 4*assay cut-off): number analyzed (Participants) | 90 | 77
  Anti-PRN, S+ (< 4*assay cut-off) | 90 | 76
  Anti-PRN, S+ (≥ 4*assay cut-off): number analyzed (Participants) | 89 | 133
  Anti-PRN, S+ (≥ 4*assay cut-off) | 86 | 133
  Anti-PRN, Overall: number analyzed (Participants) | 214 | 241
  Anti-PRN, Overall | 210 | 240

3. Secondary Outcome: Number of Seroprotected Subjects Against Anti-diphtheria, Anti-tetanus, Anti-poliovirus Type 1, Anti-poliovirus Type 2, Anti-poliovirus Type 3, Anti-HBs and Anti-PRP.
Description: Seroprotected subjects were defined as subjects with antibody concentrations/titers above or equal (≥) the assay cut-offs that are accepted immunological correlates of protection.
  0.1 IU/mL for anti-D and anti-T, 10 mIU/mL for anti-HB's, 8 ED50 for anti-polio virus (type 1,2,3) and 0.15 µg/mL for anti-PRP were considered as immunological correlates of protection.
Time Frame: Before the booster dose (Day 0)
Population: Analysis was performed on the According to Protocol (ATP) cohort for immunogenicity, which included all subjects who met eligibility criteria, received the booster dose of the study vaccines and for whom assay results were available for antibodies against at least one study vaccine antigen component, before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 223 | 244
Participants
  Anti-D | 181 | 220
  Anti-T | 215 | 232
  Anti-HBs: number analyzed (Participants) | 219 | 243
  Anti-HBs | 206 | 229
  Anti-polio 1: number analyzed (Participants) | 213 | 237
  Anti-polio 1 | 188 | 212
  Anti-polio 2: number analyzed (Participants) | 210 | 236
  Anti-polio 2 | 188 | 215
  Anti-polio 3: number analyzed (Participants) | 205 | 226
  Anti-polio 3 | 188 | 215
  Anti-PRP: number analyzed (Participants) | 222 | 244
  Anti-PRP | 161 | 166

4. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN
Description: Seropositive subjects were defined as subjects whose antibody concentration/titre was greater than or equal to the assay cut-off.
  Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti-PRN
Time Frame: Before the booster dose (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 223 | 244
Participants
  Anti-PT | 153 | 201
  Anti-FHA | 215 | 241
  Anti-PRN | 187 | 213

5. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal Serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F)
Description: Seropositive subjects were defined as subjects whose antibody concentration/titre was greater than or equal to the assay cut-off.
  Assay cut-off's for anti-pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) are 0.080 µg/mL, 0.075 µg/mL, 0.061 µg/mL, 0.198 µg/mL, 0.111 µg/mL, 0.102 µg/mL, 0.063 µg/mL, 0.66 µg/mL, 0.160 µg/mL, 0.111 µg/mL, 0.199 µg/mL, 0.163 µg/mL, 0.073 µg/mL respectively.
Time Frame: Before the booster dose (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 211 | 232
Participants
  Anti-pneumococcal serotype 1 | 196 | 214
  Anti-pneumococcal serotype 3 | 122 | 147
  Anti-pneumococcal serotype 4: number analyzed (Participants) | 209 | 232
  Anti-pneumococcal serotype 4 | 189 | 215
  Anti-pneumococcal serotype 5: number analyzed (Participants) | 211 | 229
  Anti-pneumococcal serotype 5 | 163 | 182
  Anti-pneumococcal serotype 6A | 196 | 219
  Anti-pneumococcal serotype 6B | 175 | 205
  Anti-pneumococcal serotype 7F | 210 | 232
  Anti-pneumococcal serotype 9V | 203 | 225
  Anti-pneumococcal serotype 14 | 201 | 223
  Anti-pneumococcal serotype 18C | 168 | 190
  Anti-pneumococcal serotype 19A | 148 | 172
  Anti-pneumococcal serotype 19F | 183 | 202
  Anti-pneumococcal serotype 23F: number analyzed (Participants) | 210 | 229
  Anti-pneumococcal serotype 23F | 160 | 191

6. Secondary Outcome: Anti-D, Anti-T, Anti-PT, Anti-FHA, Anti-PRN Antibody Concentrations
Description: Antibody concentrations are presented as Geometric Mean Concentrations (GMCs) and expressed in IU/mL.
Time Frame: Before the booster dose (Day 0) and One month after the booster dose (Day 30)
Population: Analysis was performed on the According to Protocol (ATP) cohort for immunogenicity, which included all subjects who met eligibility criteria, received the booster dose of the study vaccines and for whom assay results were available for antibodies against at least one study vaccine antigen component, before and after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 223 | 247
IU/ml
  Anti-D at Day 0: number analyzed (Participants) | 223 | 244
  Anti-D at Day 0 | 0.207 [0.184 to 0.234] | 0.322 [0.285 to 0.363]
  Anti-D at Day 30: number analyzed (Participants) | 221 | 247
  Anti-D at Day 30 | 6.114 [5.577 to 6.703] | 8.402 [7.694 to 9.174]
  Anti-T at Day 0: number analyzed (Participants) | 223 | 244
  Anti-T at Day 0 | 0.753 [0.646 to 0.878] | 0.578 [0.506 to 0.659]
  Anti-T at Day 30: number analyzed (Participants) | 221 | 247
  Anti-T at Day 30 | 8.200 [7.324 to 9.180] | 6.758 [6.143 to 7.433]
  Anti-PT at Day 0: number analyzed (Participants) | 223 | 244
  Anti-PT at Day 0 | 4.4 [3.8 to 5.0] | 6.3 [5.5 to 7.1]
  Anti-PT at Day 30: number analyzed (Participants) | 221 | 247
  Anti-PT at Day 30 | 52.4 [46.9 to 58.4] | 80.3 [73.3 to 88.1]
  Anti-FHA at Day 0: number analyzed (Participants) | 223 | 244
  Anti-FHA at Day 0 | 11.2 [9.6 to 13.1] | 16.5 [14.4 to 18.8]
  Anti-FHA at Day 30: number analyzed (Participants) | 221 | 247
  Anti-FHA at Day 30 | 152.5 [136.3 to 170.6] | 187.2 [172.7 to 202.9]
  Anti-PRN at Day 0: number analyzed (Participants) | 223 | 244
  Anti-PRN at Day 0 | 6.9 [5.8 to 8.2] | 9.6 [8.3 to 11.2]
  Anti-PRN at Day 30: number analyzed (Participants) | 220 | 247
  Anti-PRN at Day 30 | 333.9 [285.4 to 390.7] | 262.3 [230.9 to 298.1]

7. Secondary Outcome: Anti-poliovirus Type 1, 2, 3 Antibody Titres
Description: Anti-Poliovirus type 1, 2 and 3 antibody titers were expressed as Geometric Mean Titers (GMT).
Time Frame: Before the booster dose (Day 0) and One month after the booster dose (Day 30)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 213 | 237
Titers
  Anti-polio 1 at Day 0 | 64.9 [52.0 to 80.9] | 83.3 [67.7 to 102.5]
  Anti-polio 1 at Day 30: number analyzed (Participants) | 204 | 228
  Anti-polio 1 at Day 30 | 1611.7 [1381.2 to 1880.6] | 1532.1 [1322.2 to 1775.3]
  Anti-polio 2 at Day 0: number analyzed (Participants) | 210 | 236
  Anti-polio 2 at Day 0 | 71.7 [57.6 to 89.4] | 79.2 [64.4 to 97.5]
  Anti-polio 2 at Day 30: number analyzed (Participants) | 201 | 227
  Anti-polio 2 at Day 30 | 2232.4 [1931.2 to 2580.5] | 2371.2 [2097.9 to 2680.1]
  Anti-polio 3 at Day 0: number analyzed (Participants) | 205 | 226
  Anti-polio 3 at Day 0 | 106.0 [84.1 to 133.4] | 118.4 [97.0 to 144.5]
  Anti-polio 3 at Day 30: number analyzed (Participants) | 188 | 210
  Anti-polio 3 at Day 30 | 2944.6 [2529.4 to 3427.9] | 2891.8 [2496.2 to 3350.2]

8. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations are presented as Geometric Mean Concentrations (GMCs) and expressed in mIU/mL.
Time Frame: Before the booster dose (Day 0) and One month after the booster dose (Day 30)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 219 | 243
mIU/mL
  Anti-HBs at Day 0 | 158.7 [129.9 to 194.0] | 193.4 [158.4 to 236.1]
  Anti-HBs at Day 30: number analyzed (Participants) | 216 | 241
  Anti-HBs at Day 30 | 4858.3 [3918.4 to 6023.7] | 5031.2 [4072.7 to 6215.4]

9. Secondary Outcome: Anti-pneumococcal Serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and Anti-PRP Antibody Concentrations
Description: Antibody concentrations are presented as Geometric Mean Concentrations (GMCs) and expressed in µg/mL.
Time Frame: Before the booster dose (Day 0) and One month after the booster dose (Day 30)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 222 | 247
µg/mL
  Anti-PnPS 1 at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 1 at Day 0 | 0.22 [0.19 to 0.24] | 0.27 [0.24 to 0.30]
  Anti-PnPS 1 at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 1 at Day 30 | 3.22 [2.88 to 3.60] | 3.64 [3.28 to 4.04]
  Anti-PnPS 3 at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 3 at Day 0 | 0.08 [0.07 to 0.09] | 0.10 [0.09 to 0.11]
  Anti-PnPS 3 at Day 30: number analyzed (Participants) | 208 | 235
  Anti-PnPS 3 at Day 30 | 0.59 [0.53 to 0.65] | 0.62 [0.57 to 0.69]
  Anti-PnPS 4 at Day 0: number analyzed (Participants) | 209 | 232
  Anti-PnPS 4 at Day 0 | 0.15 [0.13 to 0.16] | 0.19 [0.17 to 0.22]
  Anti-PnPS 4 at Day 30: number analyzed (Participants) | 208 | 234
  Anti-PnPS 4 at Day 30 | 2.91 [2.54 to 3.33] | 3.28 [2.89 to 3.72]
  Anti-PnPS 5 at Day 0: number analyzed (Participants) | 211 | 229
  Anti-PnPS 5 at Day 0 | 0.33 [0.29 to 0.37] | 0.34 [0.31 to 0.38]
  Anti-PnPS 5 at Day 30: number analyzed (Participants) | 204 | 229
  Anti-PnPS 5 at Day 30 | 2.66 [2.39 to 2.97] | 2.81 [2.52 to 3.14]
  Anti-PnPS 6A at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 6A at Day 0 | 0.38 [0.33 to 0.43] | 0.44 [0.39 to 0.50]
  Anti-PnPS 6A at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 6A at Day 30 | 9.07 [8.05 to 10.22] | 9.49 [8.45 to 10.67]
  Anti-PnPS 6B at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 6B at Day 0 | 0.29 [0.25 to 0.33] | 0.33 [0.29 to 0.38]
  Anti-PnPS 6B at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 6B at Day 30 | 7.83 [6.82 to 8.98] | 8.00 [7.06 to 9.06]
  Anti-PnPS 7F at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 7F at Day 0 | 0.49 [0.44 to 0.54] | 0.56 [0.51 to 0.61]
  Anti-PnPS 7F at Day 30: number analyzed (Participants) | 208 | 235
  Anti-PnPS 7F at Day 30 | 5.00 [4.55 to 5.50] | 4.96 [4.50 to 5.48]
  Anti-PnPS 9V at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 9V at Day 0 | 0.26 [0.23 to 0.29] | 0.32 [0.28 to 0.36]
  Anti-PnPS 9V at Day 30: number analyzed (Participants) | 208 | 235
  Anti-PnPS 9V at Day 30 | 3.74 [3.35 to 4.16] | 3.91 [3.52 to 4.35]
  Anti-PnPS 14 at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 14 at Day 0 | 0.97 [0.85 to 1.11] | 1.19 [1.04 to 1.37]
  Anti-PnPS 14 at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 14 at Day 30 | 10.36 [9.22 to 11.64] | 11.62 [10.34 to 13.06]
  Anti-PnPS 18C at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 18C at Day 0 | 0.19 [0.17 to 0.21] | 0.23 [0.21 to 0.26]
  Anti-PnPS 18C at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 18C at Day 30 | 3.23 [2.86 to 3.65] | 3.57 [3.21 to 3.98]
  Anti-PnPS 19A at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 19A at Day 0 | 0.32 [0.27 to 0.37] | 0.37 [0.32 to 0.43]
  Anti-PnPS 19A at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 19A at Day 30 | 7.90 [7.06 to 8.83] | 8.68 [7.82 to 9.63]
  Anti-PnPS 19F at Day 0: number analyzed (Participants) | 211 | 232
  Anti-PnPS 19F at Day 0 | 0.37 [0.32 to 0.43] | 0.47 [0.41 to 0.55]
  Anti-PnPS 19F at Day 30: number analyzed (Participants) | 208 | 236
  Anti-PnPS 19F at Day 30 | 7.66 [6.84 to 8.57] | 8.63 [7.75 to 9.62]
  Anti-PnPS 23F at Day 0: number analyzed (Participants) | 210 | 229
  Anti-PnPS 23F at Day 0 | 0.14 [0.12 to 0.16] | 0.19 [0.16 to 0.22]
  Anti-PnPS 23F at Day 30: number analyzed (Participants) | 207 | 235
  Anti-PnPS 23F at Day 30 | 2.07 [1.83 to 2.34] | 2.38 [2.10 to 2.69]
  Anti-PRP at Day 0: number analyzed (Participants) | 222 | 244
  Anti-PRP at Day 0 | 0.371 [0.303 to 0.453] | 0.292 [0.244 to 0.349]
  Anti-PRP at Day 30: number analyzed (Participants) | 221 | 247
  Anti-PRP at Day 30 | 26.186 [22.610 to 30.327] | 19.714 [16.891 to 23.010]

10. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN.
Description: Seropositive subjects were defined as subjects whose antibody concentration/titre was greater than or equal to the assay cut-off.
  Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti- FHA and 2.187 IU/mL for anti-PRN
Time Frame: At one month after the booster dose (Day 30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 221 | 247
Participants
  Anti-PT | 220 | 247
  Anti-FHA | 221 | 247
  Anti-PRN: number analyzed (Participants) | 220 | 247
  Anti-PRN | 220 | 247

11. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness, swelling. Any redness, swelling is defined as a symptom with a surface diameter greater than 0 millimeter
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after booster vaccination of two vaccines (Infanrix hexa and Prevenar 13)
Population: The analysis was performed on the Total vaccinated cohort (TVC), which included all vaccinated subjects for whom data were available and for those with booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 257 | 275
Participants
  Pain | 134 | 154
  Redness | 143 | 169
  Swelling | 119 | 122

12. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were Drowsiness, Fever, Irritability/Fussiness and Loss of appetite.
  Fever was defined as temperature ≥37.5 degree Celsius (°C) /99.5 degree Fahrenheit (°F) for oral, axillary or tympanic route, or ≥38.0°C/100.4°F on rectal route.
Time Frame: During the 4-day (Day 0-Day 3) follow-up period after booster vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 258 | 275
Participants
  Drowsiness | 128 | 138
  Irritability | 163 | 188
  Loss of Appetite | 104 | 116
  Fever | 73 | 85

13. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day (Day 0-Day 30) follow-up period after booster vaccination
Population: The analysis was performed on the Total vaccinated cohort (TVC), which included all vaccinated subjects for whom data were available
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 263 | 277
Participants | 94 | 111

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAE is any untoward medical occurrence that results in death, is life threatening, requires hospitalisation or prolongation of existing hospitalisation, resulting in disability/incapacity
Time Frame: From booster dose up to study end (approximately 6 or 7 months, per subject)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 263 | 277
Participants | 0 | 3

15. Secondary Outcome: Number of Subjects With an ASQ-3 Score (Ages & Stages Questionnaires, Third Edition) in the Black Zone
Description: Neurodevelopmental status was measured by ASQ-3 score scale [ASQ-3, 2016] in the black zone. The ASQ-3 included a series of questions designed to assess 5 areas of development (communication, gross motor, fine motor, problem solving, and personal-social). Any subject who scored below the cut-off i.e., a score more than 2 Standard Deviations (SDs) below the mean score for the U.S. reference group (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment (using the Bayley Scale for Infant Development, Version III [BSID-III])
Time Frame: At 9 months of age, 18 months of age, and 9 or 18 months of age
Population: The analysis was performed on Total enrolled cohort, which included enrolled subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 269 | 281
Participants
  Any domain at Month 9 | 27 | 28
  Communication at Month 9 | 1 | 3
  Gross motor skills at Month 9 | 14 | 19
  Fine motor at Month 9 | 8 | 3
  Problem solving at Month 9 | 7 | 6
  Personal- Social at Month 9 | 2 | 2
  Any domain at Month 18: number analyzed (Participants) | 257 | 274
  Any domain at Month 18 | 6 | 5
  Communication at Month 18: number analyzed (Participants) | 257 | 274
  Communication at Month 18 | 1 | 0
  Gross motor skills at Month 18: number analyzed (Participants) | 257 | 274
  Gross motor skills at Month 18 | 3 | 2
  Fine motor at Month 18: number analyzed (Participants) | 257 | 274
  Fine motor at Month 18 | 1 | 1
  Problem solving at Month 18: number analyzed (Participants) | 257 | 274
  Problem solving at Month 18 | 1 | 3
  Personal- Social at Month 18: number analyzed (Participants) | 257 | 274
  Personal- Social at Month 18 | 0 | 0
  Any domain at Month 9 or 18 | 31 | 31
  Communication at Month 9 or 18 | 2 | 3
  Gross motor skills at Month 9 or 18 | 16 | 20
  Fine motor at Month 9 or 18 | 9 | 4
  Problem solving at Month 9 or 18 | 8 | 8
  Personal- Social at Month 9 or 18 | 2 | 2

16. Secondary Outcome: Number of Subjects Referred for Formal Neurodevelopmental Evaluation Using BSID-III (Bayley Scale for Infant Development, Version III)
Description: Any subject who scored below the cut-off i.e., a score more than 2 Standard Deviations (SDs) below the mean score for the U.S. reference group (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was referred to a developmental specialist for a formal neurodevelopmental assessment (using the Bayley Scale for Infant Development, Version III BSID-III)
Time Frame: At 9 months of age, 18 months of age, and 9 or 18 months of age
Population: The analysis was performed on subjects from the Total enrolled cohort, who scored, below the defined cut-off in any of the 5 domains, when using the ASQ-3 score scale.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 31 | 31
Participants
  Any Domain at Month 9: number analyzed (Participants) | 27 | 28
  Any Domain at Month 9 | 16 | 14
  Any Domain at Month 18: number analyzed (Participants) | 6 | 5
  Any Domain at Month 18 | 6 | 3
  Any Domain at Month 9 or 18 | 20 | 17

17. Secondary Outcome: Estimated Proportion of Infants With at Least One of the Indicators of Neurodevelopmental Impairment Using BSID-III (Bayley Scale for Infant Development, Version III)
Description: The estimated proportion (expressed in percentage) of infants with a BSID-III indicator of neurodevelopmental delay was based on ASQ-3 black zone indicator and subsequent BSID-III assessment using the following formula: 100 * (Number of subjects with ASQ-3 below cut off / Number of enrolled subjects with available results) * (Number of subjects with at least one indicator of neurodevelopmental delay using BSID III / Number of subjects referred for BSID III evaluation)
Time Frame: At 9 months of age, 18 months of age, and 9 or 18 months of age
Population: The analysis was performed on Total enrolled cohort, which included enrolled subjects with available results.
Measure: Number (95% Confidence Interval); unit: Percentage of Infants
Arm/Group | dTpa Group | Control Group
Number analyzed (Participants) | 269 | 281
Percentage of Infants
  Any domain at Month 9 | 4.39 [2.1 to 8.0] | 5.69 [3.0 to 9.6]
  Any domain at Month 18: number analyzed (Participants) | 257 | 274
  Any domain at Month 18 | 1.17 [0.2 to 3.4] | 0.61 [0.1 to 2.8]
  Any domain at Month 9 or 18 | 4.61 [2.3 to 8.2] | 5.84 [3.2 to 9.7]

ADVERSE EVENTS:
Time Frame: Solicited symptoms were collected during the 4-day (Day 0 - Day 3) follow-up period after each vaccination. Unsolicited AEs were collected during the 31-day (Day 0 - Day 30) follow-up period after each vaccination. SAEs were collected from booster dose up to study end (approximately 6 or 7 months, per subject)
Description: Safety analysis has been performed on the vaccinated subjects
Arm/Group | dTpa Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/277
Serious Adverse Events (participants affected / at risk) | 0/263 | 3/277
Other Adverse Events (participants affected / at risk) | 232/263 | 257/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group (N=263) | Control Group (N=277)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group (N=263) | Control Group (N=277)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 6 (6)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 4 (4) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (11) | 8 (8)
Chills (General disorders) | 1 (1) | 0 (0)
Crying (General disorders) | 2 (2) | 0 (0)
Discomfort (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 143 (143) | 169 (169)
Injection site induration (General disorders) | 1 (1) | 1 (1)
Injection site mass (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 134 (134) | 154 (154)
Injection site swelling (General disorders) | 119 (119) | 122 (122)
Pyrexia (General disorders) | 81 (85) | 101 (109)
Vaccination site irritation (General disorders) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5) | 6 (6)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Candida nappy (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 9 (9) | 5 (5)
Croup infectious (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 9 (9) | 12 (13)
Exanthema subitum (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 5 (5)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 2 (2)
Herpangina (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 4 (4) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 12 (13) | 10 (11)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (4) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (5) | 5 (6)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 3 (3)
Roseola (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 4 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 9 (9)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 3 (3)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 104 (104) | 116 (116)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mastocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 128 (128) | 138 (138)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 163 (164) | 189 (191)
Genital erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02853929/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT02853929/SAP_001.pdf